CLINICAL TRIAL: NCT06140498
Title: Effects of Self-Efficacy Ecological Momentary Intervention (EMA) App
Acronym: EMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The New School (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Adam Brown, Ph.D., Associate Professor of Psychology (Clinical) and Vice Provost for Research, The New School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-96
Record Dates: First submitted 2023-09-11; First posted 2023-11-20 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-08

CONDITIONS: Self Efficacy
MeSH Terms: interventions — Ecological Momentary Assessment

STUDY DESIGN:
Intervention Model Description: Random Allocation, 2 Arms allocation to groups blinded, parallel assignment, masking participant, outcome assessor, investigator.
Who Masked: Investigator
Masking Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Digital Self-Efficacy Training with 3 trainings daily and Ecological Momentary Assessment
  Interventions: Behavioral: Self-Efficacy Training and Ecological Momentary Assessment
- Control (Active Comparator): Ecological Momentary Assessment
  Interventions: Behavioral: Control intervention: Ecological Momentary Assessment only

INTERVENTIONS:
Behavioral: Self-Efficacy Training and Ecological Momentary Assessment — Participants receive 3 self-efficacy trainings per day, combined with Ecological Momentary Assessments assessing mood, social contacts, and virtual context 3x/day for one week
  Arms: Intervention
Behavioral: Control intervention: Ecological Momentary Assessment only — Participants receive Ecological Momentary Assessments assessing mood, social contacts, and virtual context 3x/day for one week only
  Arms: Control

SUMMARY:
This "SeApp" study aims to test a self-efficacy Ecological Momentary Intervention (EMI) in healthy students in the context of COVID-19. EMIs are mostly smartphone-based applications that deliver interventions to people while being engaged in their daily life activities. The app harnesses the power of self-efficacy autobiographical memories (e.g. problem-solving memories, memories of success).

Ecological Momentary Assessments (EMAs) are also incorporated into the study to capture individuals' feelings, affect, and behavior in real time.

Clarification added [September 2025]: The record previously showed an incorrect estimated enrollment due to a data entry error. The planned enrollment for this trial was 93, consistent with comparable prior studies, and enrollment was closed when 93 participants had been enrolled.

DETAILED DESCRIPTION:
This "SeApp" study aims to test a self-efficacy Ecological Momentary Intervention (EMI) in healthy students in the context of COVID-19. EMIs are mostly smartphone-based applications that deliver interventions to people while being engaged in their daily life activities. The app harnesses the power of self-efficacy autobiographical memories (e.g. problem-solving memories, memories of success).

Ecological Momentary Assessments (EMAs) are also incorporated into the study to capture individuals' feelings, affect, and behavior in real time.

Developed by psychologist Dr. Albert Bandura in 1977, the concept of self-efficacy refers to an individual's belief in their ability to perform the necessary actions to manage particular situations. Bandura's theory highlights four major components of self-efficacy, including mastery experiences, socialmodeling, social persuasion, and psychological responses. The app tested here focuses on mastery experiences, which are what individuals gain when they take on a challenge and succeed. The app prompts participants in the daily recall of self-efficacy memories. The project aims to test its feasibility and to investigate how daily self-efficacy and motivation can be enhanced and perceived stress and depression reduced by daily memory-based training via smartphone app.

ELIGIBILITY:
Inclusion Criteria:

1. Value on Perceived Stress Scale ≥ 13
2. Student
3. Owner of a smartphone

Exclusion Criteria:

1. Psychiatric history

-

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
General Self-Efficacy | after app completion and 1 month after app completion
  change in general self-efficacy meeasured using the General Self-Efficacy Scale (GSE, 10 items rated on a 4-point Likert scale with higher scores indicating greater levels of self-efficacy; min=10, max=40)

SECONDARY OUTCOMES:
Perceived Stress | after app completion and 1 month after app completion
  change in perceived stress measured using the Perceived Stress Scale (PSS; 10 items rated on a 0-4 scale with higher scores indicating greater levels of perceived stress; min=0, max=40)
Intolerance of Uncertainty | after app completion and 1 month after app completion
  change in intolerance of uncertainty measured using the Intolerance of Uncertainty Scale (IUS; 12 items rated on a 5-point Likert scale with higher scores indicating greater intolerance of uncertainty; min=12, max=60)
State and Trait Anxiety | after app completion and 1 month after app completion
  change in state and trait anxiety measured using the The State-Trait Anxiety Inventory (STAI; 40 items rated on a 4-point Likert scale with a commonly used cutoff score of 40 indicating probable clinical levels of anxiety; min=20, max=80 on the subscales)
Positive and Negative Affect positive and negative affect | after app completion and 1 month after app completion
  change in positive and negative affect measured using the Positive and Negative Affect Scale (PANAS; 20 items rated on a 5-point Likert scale with 10 items measuring positive affect and 10 items measuring and higher scores indicating greater levels of positive or negative affect; min=10, max=50 on the subscales)
Hopelessness | after app completion and 1 month after app completion
  change in hopelessness measured using the BHS
Depression | after app completion and 1 month after app completion
  change in depression measured using the Beck Hopelessness Scale (BDI-II; 20 true and false items with higher scores indicating greater levels of hopelessness)

OTHER OUTCOMES:
Ecological Momentary Assessment | through app participation (1 week)
  change of momentary mood
Hope | after app completion and 1 month after app completion
  change in hope measured using the Adult Hope Scale (AHS; consists of 12 items, and respondents are required to rate each item on an 8-point Likert scale; min=12, max=96)
Satisfaction with Mobile Application | single time point: immediately after the intervention
  to evaluate usage of app using the User version of the Mobile Application Rating Scale (uMARS; consists of 20 itesm, scores ranges from 1 to 5; the total score could range from 20 to 100, with higher scores indicating a higher overall quality rating for the app)
Coronavirus Anxiety Scale | after app completion and 1 month after app completion
  to evaluate association with coronoavirus anxiety the coronavirus anxiety scale is used (10 items, each rated on a scale of 0 to 4, the total score could range from 0 to 40)
Self-efficacy memories | single time point: baseline
  exploratory (descriptive) analysis, using no scale

CONTACTS AND LOCATIONS:
Locations (1):
- The New School, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No